CLINICAL TRIAL: NCT02892058
Title: Development of a Tool for the Self-assessment of Flare in Patients With Osteoarthritis of Lower Limbs
Brief Title: Self-assessment of Flare in Osteoarthritis of Lower Limbs
Acronym: FLARE-OA
Status: Completed | Type: Observational
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, GUILLEMIN Francis, MD, Professor, Central Hospital, Nancy, France
Other Study IDs: FLARE-OA
Record Dates: First submitted 2016-08-23; First posted 2016-09-08 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Osteoarthritis
MeSH Terms: conditions — Osteoarthritis

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The need for a tool to measure flare in lower limb osteoarthritis (OA of the hip and knee) is justified by the opportunities for development of clinical trials targeting hip and knee OA long-term treatment (slow acting drug, disease modifying drug) and short-term treatment of symptoms. Such treatments are currently under development and will likely bring important changes in the treatment of patients. The development of a Flare-OA tool would be essential to capture the occurrence of flare, and to implement and adapt treatment strategies.

This project was elaborated with the aims to:

1. define the construct through development of a conceptual framework
2. use the conceptual framework to inform the development of a patient-reported outcome measure, Flare-OA tool, for people with OA
3. evaluate the psychometric properties of the new measure using the OMERACT (Outcome Measures in Rheumatology) filter 2.0 and Rasch measurement methods.

DETAILED DESCRIPTION:
Chronologically, the development of a Flare-OA (osteoarthritis) tool will be addressed in the first part of the project (Part 1) and its psychometric validity was evaluated in the second part (Part 2).

Part 1 of the project: The development of the Flare-OA tool will be conducted in several steps, and needs multiple proficiencies in qualitative research (health psychologist), in quantitative research (epidemiologist, psychometrician), in experience of the disease (patients), and in experience of care of the disease (health care professionals).

Two approaches will be taken to define the construct of a flare in lower limb OA: A review of the literature, and the development of a conceptual framework informed by the results of the literature. To help define/conceptualize the construct "Flare in OA" a procedure will be implemented to identify (what are the key variables, or symptoms, that get worse) and clarify (how exactly these variables are described in the literature, by patients, and by clinicians.

Participants :

1. - Patients should be representative of the disease spectrum, i.e. of prevalent cases. They will be recruited in clinical settings and epidemiological sources.
2. - Health care professionals (HCP) will include General Practitioners, Rheumatologists, Rehabilitation specialists, Orthopaedic surgeons, Nurse in general practice or orthopedic wards, Physiotherapists.

ELIGIBILITY:
Inclusion Criteria:

* with clinical and radiological hip or knee OA confirmed by a physician,
* whatever their status regarding flare of OA. The intention of the Flare-OA tool is not to detect current flare only, but also a flare that may have occurred before the encounter with the health care professional. Therefore patient will not be selected on flare, and patients with flare will not be excluded.

Exclusion Criteria:

* Patients who never experienced nor currently report having a flare of OA
* Patients with both hip and knee OA

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with knee or hip osteoarthritis (OA).
  France: several sources will be sollicited including:
  * investigators in rheumatology and general practitioner network in each participating centre,
  * Patients participating in the KHOALA cohort, a representative prevalent case cohort study followed-up in 6 centres.
  Australia: patients participating in the online cohort SPARK-web study Canada : patients will be recruited in Toronto osteoarthritis center.
Sampling Method: Non-Probability Sample
Enrollment: 398 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2022-12 (Actual); Study Completion 2022-12 (Actual)

PRIMARY OUTCOMES:
Ability of a FLARE-OA self-questionnaire to detect flare episodes in knee or hip osteoarthritis | Baseline
  patient-reported outcome questionnaire for the self-assessment of flare in osteoarthritis. The questionnaire will be developed during the first part of the study.
Change in ability of a FLARE-OA self-questionnaire to detect flare episodes in knee or hip osteoarthritis during a 6 months period | At 3 and 6 month follow-up
  patient-reported outcome questionnaire for the self-assessment of flare in osteoarthritis. The questionnaire will be developed during the first part of the study.

SECONDARY OUTCOMES:
Evolution of the quality of life during a 6 months period with the standardized OAKHQOL questionnaire | up to 3 and 6 month
  Osteoarthritis knee and hip quality of life questionnaire (OAKHQOL) self-assessment questionnaire
Evolution of the functional limitation related to knee osteoarthritis during a 6 months period with the standardized KOOS questionnaire | up to 3 and 6 month
  Knee injury and Osteoarthritis Outcome Score (KOOS) patient questionnaire. Standardized answer options are given (5 Likert boxes) and each question is assigned a score from 0 to 4.
Evolution of the functional limitation related to hip osteoarthritis during a 6 months period with the standardized HOOS questionnaire | up to 3 and 6 month
  Hip disability and Osteoarthritis Outcome Score (HOOS) patient questionnaire. Standardized answer options are given (5 Likert boxes) and each question gets a score from 0 to 4.
Pain intensity measure | up to 3 and 6 month
  Self-reported pain intensity using a numerical rating scale

CONTACTS AND LOCATIONS:
Overall Officials: Francis GUILLEMIN, Principal Investigator — CHRU NANCY, CIC 1433 Epidémiologie Clinique
Locations (12):
- Institute of Bone and Joint Research - University of Sydney, Sydney, Australia
- University of Toronto, Toronto, Canada
- France (9):
  - CHU Jean Minjoz, Besançon
  - CHU La Cavale Blanche, Brest
  - CHU Hôpital Général, Dijon
  - CHU Hôpital Sud A. Michallon, Grenoble
  - CHRU Hôtel Dieu, Nantes
  - AP-HP Saint Antoine, Paris
  - AP-HP La Pitié, Paris
  - CHU de Poitiers, Poitiers
  - CHRU, Rhumatologie, Vandœuvre-lès-Nancy
- CHU Fort de France, Fort-de-France, Martinique

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] King LK, Epstein J, Cross M, Buzzi M, Buttel T, Cembalo SM, Spitz E, Adams CL, Adebajo A, Bennell K, Blanco B, Courage U, Decary S, Gill M, Gill TK, Hajji R, Hinman RS, Jones A, Li LC, Mather K, Mani R, Nasef SI, Oo WM, Osteras N, Otobo TM, Ramiro S, Sharma S, April KT, Touma Z, Whittaker JL, Wluka AE, Grosskleg S, Hunter DJ, Shea B, Hawker GA, Callahan LF, March L, Guillemin F. Endorsement of the domains of knee and hip osteoarthritis (OA) flare: A report from the OMERACT 2020 inaugural virtual consensus vote from the flares in OA working group. Semin Arthritis Rheum. 2021 Jun;51(3):618-622. doi: 10.1016/j.semarthrit.2021.03.010. Epub 2021 Mar 20. PMID 33775461
- [Result] Guillemin F, Ricatte C, Barcenilla-Wong A, Schoumacker A, Cross M, Alleyrat C, Buttel T, Cembalo M, Manseur H, Urban H, Fautrel B, Conaghan PG, Hawker G, Rutherford C, March L, Spitz E, Hunter DJ. Developing a Preliminary Definition and Domains of Flare in Knee and Hip Osteoarthritis (OA): Consensus Building of the Flare-in-OA OMERACT Group. J Rheumatol. 2019 Sep;46(9):1188-1191. doi: 10.3899/jrheum.181085. Epub 2019 May 15. PMID 31092709
- [Result] Traore Y, Epstein J, Spitz E, March L, Maillefert JF, Rutherford C, Ricatte C, Alleyrat C, Cross M, King LK, Callahan LF, Fautrel B, Buttel T, Hawker G, Hunter DJ, Guillemin F. Development and validation of the Flare-OA questionnaire for measuring flare in knee and hip osteoarthritis. Osteoarthritis Cartilage. 2022 May;30(5):689-696. doi: 10.1016/j.joca.2021.12.011. Epub 2022 Jan 20. PMID 35066175